CLINICAL TRIAL: NCT05940246
Title: The Empowerment Study
Brief Title: Investigating the Role of Motivational Interviewing in Swedish Patients Undergoing Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The Empowerment TKA Study
Record Dates: First submitted 2023-06-20; First posted 2023-07-11 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee arthroplasty; Patient empowerment; Motivational interviewing
MeSH Terms: conditions — Osteoarthritis, Knee; Patient Participation | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing (Experimental): Motivational Interviewing over the phone 1 time before surgery and 6 times (3-5 weeks interval) the first 6 months after surgery. Patients can contact a physical therapist in the first 6 months after surgery for additional questions and extra support.
  Interventions: Behavioral: Motivational Interviewing
- Standard treatment (No Intervention): Standard treatment

INTERVENTIONS:
Behavioral: Motivational Interviewing — MI was introduced by William Miller in 1983 as a strategy to promote behavioral changes that would make people drink less. It is well established that MI can be successfully applied to many areas across the medical disciplines. Although the aim of MI is behavioral changes toward a specific goal it is necessary to understand the essence of MI with the "four key interrelated elements of the spirits of MI". These are partnership, acceptance, compassion, and evocation. Together they form an equal and respectful collaboration between the MI practitioner and the patient wherein empathy and acknowledgment are important pillars. Moreover, an important message derived from the spirit of MI is the belief that patients in themselves have and know what is needed and get support from the MI practitioner to find it.
  Arms: Motivational interviewing

SUMMARY:
Knee arthroplasty is a successful surgical treatment for end-stage osteoarthritis. Most patients are satisfied with the result, however, 10% of the patients have remained dissatisfied over the last decades despite the advantages of the surgical procedure. Previous studies suggest that rehabilitation needs to be individualized and that some patients request additional support.

Patient empowerment is a patient-centered strategy to increase, amongst other, patient engagement, participation, and motivation. Patient empowerment can be defined as a "process that helps people gain control over their own lives and increases their capacity to act on issues that they themselves define as important". One way of increasing patient empowerment is through motivational interviewing. Motivational interviewing is an evidence-based approach in which patients are supported to identify behavior changes toward their own individual goals.

The aim of this study is to investigate if motivational interviewing could increase satisfaction in patients undergoing knee arthroplasty. Furthermore, we want to examine role MI in this patient group with interviews of both MI-practitioners and patients as well as detailed investigations about the MI sessions.

ELIGIBILITY:
Inclusion Criteria:

Scheduled for primary knee arthroplasty

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the rehabilitation | Assessed 6 months postoperatively
  Patient reported outcome. Question: "How would you define your level of satisfaction with the rehabilitation?" Answer options: (1) Very satisfied, (2) Satisfied, (3) Neither, (4) Dissatisfied and (5) Very dissatisfied
Satisfaction with the rehabilitation | Assessed 12 months postoperatively
  Patient reported outcome. Question: "How would you define your level of satisfaction with the rehabilitation?" Answer options: (1) Very satisfied, (2) Satisfied, (3) Neither, (4) Dissatisfied and (5) Very dissatisfied
Satisfaction with the knee | Assessed 6 months postoperatively
  Patient reported outcome. Question: "How would you define your level of satisfaction with your operated knee?" Answer options: (1) Very satisfied, (2) Satisfied, (3) Neither, (4) Dissatisfied and (5) Very dissatisfied
Satisfaction with the knee | Assessed 12 months postoperatively
  Patient reported outcome. Question: "How would you define your level of satisfaction with your operated knee?" Answer options: (1) Very satisfied, (2) Satisfied, (3) Neither, (4) Dissatisfied and (5) Very dissatisfied

SECONDARY OUTCOMES:
Knee awareness | Preoperatively, 6 months postoperatively and 12 months postoperatively
  Assessed by the Forgotten Joint Score-12 (FJS)
Self-reported pain and function | Preoperatively, 6 months postoperatively and 12 months postoperatively
  Assessed by the Knee Injury and Osteoarthritis Outcome Score (KOOS)
Knee function | Preoperatively, 6 months postoperatively and 12 months postoperatively
  Assessed by the "5 times sit to stand"-test. Patients receive written instructions and perform the test themselves at home.
Patient reported experience measures | 12 months postoperatively
  Three questions own patients own experiences
  1. "Did you receive the support you expected after your knee surgery?" Answer options: (1) Yes, more support than expected, (2) Yes, as much support as expected, (3) No, less support than expected and (4) No, considerably less support than expected
  2. "Did you participate in and had influence over the rehabilitation as you expected?" Answer options: (1) Yes, to very high degree, (2) Yes, to a high degree, (3) No, less than expected and (4) No, more than I wished for
  3. "Were you treated with dignity and respect in the contacts concerning your knee surgery from after the surgery until today" Answer options: (1) Yes, to a very high degree, (2) Yes, to a high degree, (3) No, to a low degree and (4) No, not at all
Knee improvement | 6 months postoperatively, 12 months postoperatively
  Patient reported outcome. "Has your knee improved from the surgery?" Answer options: (1) Yes, the knee improved a lot from the surgery, (2) Yes, the knee improved a little bit from the surgery, (3) The surgery made no difference on the knee, (4) No, the knee is a little worse after surgery and (5) No, the knee is a lot worse after surgery

OTHER OUTCOMES:
Depression | Preoperatively, 6 months postoperatively and 12 months postoperatively
  Assessed by the Patient Health Questionnaire-9 (PHQ-9)
Health related quality of life | Preoperatively, 6 months postoperatively and 12 months postoperatively
  Assessed by the Short Form Health Survey (SF-36)
Expectations on the rehabilitation | Preoperatively
  Patient reported outcome. Question: "How would you define your expectations on the rehabilitation?" Answer options: (1) Very high, (2) High, (3) Neither, (4) Low and (5) Very low
Expectations on the surgical result | Preoperatively
  Patient reported outcome. Question: "How would you define your expectations on the final surgical result?" Answer options: (1) Very high, (2) High, (3) Neither, (4) Low and (5) Very low
Recordings of MI | 0 to 6 months postoperatively
  All 6 postoperative MI-calls on all patients in the intervention group is recorded and will be analysed by a group (MIQA-gruppen) that specialises in coding MI-calls.

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Hedström, Professor, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Capio Ortopediska Huset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided